CLINICAL TRIAL: NCT04463420
Title: Safety and Efficacy of PHR 160 Spray on the Outcomes of Patients With COVID-19 a Multi-center Randomized Blinding Clinical Trial Study
Brief Title: Safety and Efficacy of PHR 160 Spray on the Outcomes of Patients With COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baqiyatallah Medical Sciences University (Other)
Responsible Party: Principal Investigator, Mohammad Sadegh Bagheri Baghdasht, Principal Investigator, Baqiyatallah Medical Sciences University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IR.BMSU.REC.1399.176
Record Dates: First submitted 2020-07-04; First posted 2020-07-09 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Intervention group: : Hydroxychloroquine 400 mg only on the first day / one naproxen 250 mg every 12 hours for 5 days / 500 mg azithromycin on the first day and 250 mg on the second to fifth days / 40 mg famotidine every 12 hours for 5 days / 25 mg prednisolone daily for 5 days / PHR160 spray one hour oral puff with Demyar ten times a day for ten days in a row, for ten days.
  Interventions: Drug: PHR160 Spray; Drug: Standard treatment
- Control Group (Placebo Comparator): Control group: Hydroxychloroquine 400 mg only on the first day / one naproxen 250 mg every 12 hours for 5 days / 500 mg azithromycin on the first day and 250 mg on the second to fifth days / 40 mg famotidine every 12 hours for 5 days Daily / 25 mg prednisolone daily for 5 days / placebo spray one hourly oral puff ten times a day for ten days in a row, for ten days
  Interventions: Drug: Placebo; Drug: Standard treatment

INTERVENTIONS:
Drug: PHR160 Spray — One puff spray per hour containing 300 mg of the drug will be given to patients. This treatment lasts up to 10 days.
  Arms: Test Group
Drug: Placebo — participants will receive a placebo spray every hour. This process will continue for 10 days.
  Arms: Control Group
Drug: Standard treatment — : Hydroxychloroquine 400 mg only on the first day / one naproxen 250 mg every 12 hours for 5 days / 500 mg azithromycin on the first day and 250 mg on the second to fifth days / 40 mg famotidine every 12 hours for 5 days / 25 mg prednisolone daily for 5 days

SUMMARY:
This study is a multi-center randomized, controlled, and blinded clinical trial study that will be performed in four medical-educational centers. In this study, the samples will be selected from among patients with SARS-CoV-2 as easy access and based on entry criteria and will be randomly divided into two groups, including a control group and an intervention group. The study will be conducted in four medical centers. From each center, 56 definitive Corona patients will be selected, who will be randomly divided into two groups of 28, for a total of 224 patients will enter the study. In the intervention group, in addition to receiving the test spray, Patients will also receive standard treatment

ELIGIBILITY:
Inclusion Criteria:

* Conscious consent to participate in the study
* Patients 18 to 75 years of age with COVID-19 who have been diagnosed with PCR.
* Strong clinical suspicion of covid 19 with positive findings in CT Scan
* Shortness of breath

Exclusion Criteria:

* Patients with HIV
* Patients with cancer undergoing chemotherapy
* Patients receiving Immune Mediators
* Patients need hospitalization in the intensive care unit
* Patients with uncontrolled heart, kidney or liver failure
* Pregnant or lactating women
* Intolerance to the drugs used in this study (symptoms such as diarrhea, nausea, vomiting and respiratory problems)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2020-11-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Dyspnea | up to 14 days
  shortness of breath measured by Visual analog scale (VAS) dyspnea score. The minimum score is zero means shortness of breath and the highest score is 10 means the maximum intensity of shortness of breath.

SECONDARY OUTCOMES:
long of hospitalization | up to 28 days
  The length of time the patient is hospitalized after the diagnosis of COVID-19
Radiological Treatment Response | up to 14 days
  CT scans help determine how much the lungs are affected by COVID-19.
Mortality | Up to 28 days
  In-hospital mortality
Allergic drug | up to 14 days
  There will be known allergic reactions to the drugs.
Laboratory Treatment Response | up to 14 days
  Normal blood cell count and CRP count (normal laboratory range)
O2 saturation without supplemental oxygen | up to 14 days
  Using an oximeter pulse, the amount of oxygen saturation is measured. If the patient is receiving oxygen, first cut off the oxygen for 5 minutes and then measure. If the oxygen drops below 90 degrees, oxygen therapy will be re-established immediately.
drug reactions Adverse | Up to 14 days
  Complications in both groups should be evaluated and evaluated during treatment.
  protective response that serves to clear the trachea, bronchi, and/or lungs of irritants and secretions that measured by Physical examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammad Sadegh Bagheri Baghdasht, Tehran, Iran